CLINICAL TRIAL: NCT06084533
Title: CS1P1 PET Studies of Neuroinflammation in Parkinson Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202306067
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson Disease
  Interventions: Drug: [11C]-CS1P1
- Healthy Control
  Interventions: Drug: [11C]-CS1P1

INTERVENTIONS:
Drug: [11C]-CS1P1 — Participants will receive a single intravenous bolus injection of 10.0 - 20.0 milliCurie (mCi) of the investigational radiotracer [11C]-CS1P1. Participants will then undergo a [11C]-CS1P1 PET scan.

SUMMARY:
Parkinson disease (PD) is a progressive neurological disorder strongly linked to advancing age that results in decline in mobility and thinking. Based on prior research, the investigators think that small amounts of inflammation in the brain may contribute to the mobility and thinking problems in people with PD. They are trying to measure inflammation in the brain in order to understand how this inflammation could be contributing to the symptoms of PD. This study involves a brain positron emission tomography (PET) scan with a new, investigational radioactive tracer called [11C]-CS1P1 to identify inflammation in the brain.The goal of this project is to quantify neuroinflammation with [11C]-CS1P1 PET and compare to motor and cognitive function in participants with various stages of severity of PD compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson Disease (PD) participants must be at least 50 years old and meet clinical diagnostic criteria of idiopathic PD.
* Control participants must be at least 50 years old and not have PD, no first-degree family member with PD, and no evidence of PD or dementia on examination.

Exclusion Criteria:

* any history of other neurologic illness (e.g. stroke, seizure, multiple sclerosis)
* history of brain surgery or major head trauma
* major medical/systemic illness
* severe psychiatric illness (e.g. bipolar disorder, schizophrenia)
* major drug abuse
* history of long term use of anti-dopaminergic medication
* chronic treatment with immunomodulatory or anti-inflammatory medications
* weight over 300 lbs
* contraindication to or inability to tolerate MRI

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 50 participants with idiopathic PD and up to 30 healthy control participants are to be studied. Some of these participants will be recruited from existing research studies. Others will be recruited from the clinic, the community, and a registry of healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
PET imaging studies of [11C]-CS1P1 in healthy control participants and participants with Parkinson Disease. | At the time of PET scan
  The investigators hypothesize that specific binding of [11C]-CS1P1 is elevated in participants with neurodegenerative disease of the central nervous system compared to healthy control participants.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L White, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States